CLINICAL TRIAL: NCT00774241
Title: An Open Label Study of the Effect of First Line Combination Treatment With Avastin and Docetaxel on Disease Response in Patients With Metastatic Breast Cancer
Brief Title: PRIMADOS Study:A Study of Avastin (Bevacizumab) Plus Docetaxel for First Line Treatment of Patients With Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was put on hold then out of Medical Plan therefore cancelled
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21343
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: docetaxel

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv every 3 weeks
Drug: docetaxel — 75mg/m2 every 3 weeks for 18 weeks

SUMMARY:
This single arm study will assess the efficacy and safety of first line combination treatment with Avastin + docetaxel in patients with HER2 negative metastatic breast cancer.Patients will receive Avastin (15mg/kg iv every 3 weeks) plus docetaxel (75mg/m2 every 3 weeks for 6 cycles). The anticipated time on study treatment is until disease progression, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients, >=18 years of age;
* stage IV, HER2 negative metastatic breast cancer;
* candidate for taxane-based therapy;
* ECOG performance status 0-2.

Exclusion Criteria:

* prior chemotherapy for metastatic breast cancer;
* concomitant primary malignant disease, except for adequately treated cervical cancer in situ, or basal or squamous cell skin cancer within last 5 years;
* suspicion of CNS metastasis;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Response rate, median progression free survival, overall survival | Event driven

SECONDARY OUTCOMES:
Adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche